CLINICAL TRIAL: NCT01529099
Title: A Prospective, Non-comparative, Single Centre Study to Determine the Performance & Survivorship of the SIGMA HP® PARTIAL KNEE SYSTEM.
Brief Title: Postmarketing Study to Determine Performance of the SIGMA HP® PARTIAL KNEE SYSTEM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT10/01
Record Dates: First submitted 2011-12-06; First posted 2012-02-08 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2015-06

CONDITIONS: Osteoarthritis; Post-traumatic Arthritis; Gout; Pseudo-gout
Keywords: Osteoarthritis; Knee; Knee replacement; Knee implant; Knee arthroplasty; Unicompartmental; Primary; Partial; Patellofemoral; Medial; Lateral; Bicompartmental; Cemented; Post-traumatic arthritis of the tibio-femoral and/or patellofemoral articular surfaces; History of Gout or pseudo-gout.
MeSH Terms: conditions — Osteoarthritis; Gout; Chondrocalcinosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sigma HP Partial Knee (Experimental): Partial knee replacement
  Interventions: Device: SIGMA HP PARTIAL KNEE

INTERVENTIONS:
Device: SIGMA HP PARTIAL KNEE — SIGMA HP PARTIAL KNEE
  Other Names: Sigma HP Partial Knee Femoral component; Sigma HP Partial Knee Tibial component; Sigma HP Partial Knee Tibial insert component; Sigma Patellae; Sigma HP Partial Knee Trochlear component

SUMMARY:
This is a postmarketing study to assess the overall performance and survivorship of the SIGMA HP® PARTIAL KNEE SYSTEM.

DETAILED DESCRIPTION:
The purpose of this study is to collect more information about the Sigma HP® Partial Knee System made by DePuy International. The aim of this study is to measure how this particular type of knee replacement performs over a two year period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged at least 21 years.
* Subjects who are able to give voluntary, written informed consent to participate in this clinical investigation and from whom consent has been obtained.
* Subjects, who, in the opinion of the Clinical Investigator, are able to understand this clinical investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.
* Subject has non-inflammatory degenerative joint disease (NIDJD), including: osteoarthritis, posttraumatic arthritis, avascular necrosis and chondrocalcinosis.
* Subject has a functional stable knee.
* Subject, in the opinion of the Investigator, is suitable for either a single or bicompartmental knee replacement.
* Subject meets the following selected radiographic parameters:

  * X-ray evaluation confirms the presence of NIDJD
  * Disease location: 1 to 2 compartments, maximum. Disease can be present in the patellofemoral compartment, the medial tibiofemoral compartment, lateral tibiofemoral compartments alone or in any two compartments.
  * Disease severity: Kellgren and Lawrence44 Grade II or greater for all compartments replaced.

Exclusion Criteria:

* Subjects who, in the opinion of the Clinical Investigator, have an existing condition that would compromise their participation and follow-up in this clinical investigation.
* Women who are pregnant.
* Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.
* Subjects who have participated in a clinical investigation with an investigational product in the last 3 months.
* Subjects who are currently involved in any injury litigation claims.
* Multiple joint involvement that will compromise rehabilitation (for example: advanced hip, ankle or spine disease).
* Known to be a prisoner, mentally incompetent, an alcohol / drug abuser, involved in medical-legal case or worker's compensation
* Previous knee arthroplasty (any type) in any one of the three compartments of the knee.
* Requires more than a lateral soft tissue release or an anterior cruciate ligament reconstruction.
* Uncorrectable anatomical tibio-femoral angle.
* Bone deficiency requiring structural bone grafts to support the implants.
* Previous patellectomy.
* For Subjects indicated for a patellofemoral arthroplasty, Subject has uncorrected patella baja (Caton-Deschamps ratio less than or equal to 0.6).
* Tri-compartmental disease process (patella-femoral, medial tibio-femoral and lateral tibio-femoral).
* Active bacterial infection that may spread to other areas of the body (e.g., osteomyelitis, pyogenic infection of knee joint, urinary tract infection, etc.).
* Significant neurological or musculoskeletal deformity or a disease that may affect gait or weight bearing, (e.g., muscular dystrophy, multiple sclerosis, amputation).
* Known allergy to implant materials.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-01; Primary Completion 2015-01 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Survivorship (revision) | 2 years
  Kaplan Meier Survival analysis at 2 years (based on revision of the femoral or tibial components)

OTHER OUTCOMES:
Types and Frequency of Adverse Events | Throughout the study
Clinical outcome using the AKS score | 6 weeks, 6 months, 1 year and 2 years post-op
Patient-reported outcome using the KOOS assessment | 6 weeks, 6 months, 1 year and 2 years post-op
Patient-reported outcome using the HAAS assessment | 6 weeks, 6 months, 1 year and 2 years post-op
Patient-reported outcome using the Kujala score | 6 weeks, 6 months, 1 year and 2 years post-op
Patient-reported outcome using the Oxford Knee Score | 6 weeks, 6 months, 1 year and 2 years post-op
Patient-reported outcome using the EQ-5D assessment | 6 weeks, 6 months, 1 year and 2 years post-op
Radiographic assessment | 6 weeks, 6 months, 1 year and 2 years post-op

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (2):
  - Orthopedic Institute IRCCS Galeazzi, Milan
  - CDC, Citta di Palma, Parma
- Schulthess Klinik, Zurich, Switzerland